CLINICAL TRIAL: NCT03532893
Title: Predictive Value of Combining Inflammatory Biomarkers and Rapid Decline of FEV1 for COPD in Chinese Population - a Prospective Cohort Study
Brief Title: Predictive Value of Inflammatory Biomarkers and FEV1 for COPD
Acronym: PIFCOPD
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Collaborators: The Second Hospital of Hebei Medical University (Other); Henan Provincial People's Hospital (Other); Second Hospital of Jilin University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Shandong Provincial Hospital (Other Government); Shanxi Dayi Hospital (Other); Tianjin Medical University General Hospital (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Principal Investigator, Guangfa Wang, Head of Respiratory and critical Medicine, Principal Investigator, Clinical Professor, Peking University First Hospital
Other Study IDs: 2017YFC1309500-1
Record Dates: First submitted 2018-03-29; First posted 2018-05-22 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: COPD; FEV1
Keywords: COPD incidence; Decline in FEV1; Inflammatory biomarkers; EBC; microRNA-23a
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma，whole blood，exhaled breath condensate
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — This is a multi-center,observational, prospective, cohort study. A total of 10,000 subjects aged 40～75 without history of lung disease will be recruited and followed for 3 years. So there is no intervention in this study.

SUMMARY:
This is a multi-center, prospective, cohort study. A total of 10,000 people aged 40～75 without lung disease will be recruited and followed for 3 years. By measure the rate of decline in forced expiratory volume at one second（FEV1） and baseline inflammatory biomarkers in exhaled breath condensate and peripheral blood, we aim to explore the predictive model for chronic obstructive pulmonary disease（COPD） in China.

DETAILED DESCRIPTION:
This is a multi-center, prospective, cohort study. A total of 10,000 subjects aged 40～75 without history of lung disease will be recruited and followed for 3 years. The Department of Respiratory and Critical Care of Peking University First Hospital is responsible for this research. Other 9 units participating in the study, include the The Second Hospital of Hebei Medical University, Henan Provincial People's Hospital, The Second Hospital of Jilin University, The First Affiliated Hospital of Xi'an Jiaotong University, Shandong Provincial Hospital Affiliated to Shandong University,Shanxi Dayi Hospital, Tianjin Medical University General Hospital, The Affiliated Hospital of Inner Mongolia Medical University,The First Hospital of Qinhuangdao. Some questionnaire such as St George's Respiratory Questionnaire (SGRQ), income class, educational level, comorbidity, smoking habit and biomass smoke exposure history will be collected. The baseline level of Interleukin 6 (IL-6), high-sensitivity C-reactive Protein (hs-CRP), microRNAs-23a (miR-23a) in peripheral blood and pH value in exhaled breath condensate (EBC) will be measured, lung spirometry will be tested in the first, second and fourth years. Primary outcome is the incidence of COPD, multivariate regression analysis will be used to establish the predictive model for COPD in China.

The study protocol has been approved by the Peking University First Hospital Institutional Review Board (IRB) (2018-31). Any protocol modifications will be submitted for the IRB review and approval.

ELIGIBILITY:
Inclusion Criteria:

1. aged at 40-75 years old;
2. FEV1/FVC>70% after inhaled bronchodilator
3. have willing to participate in this study, follow the research program and have the ability to sign the informed consent;
4. lived in a community for more than 1 years and has no plans to move out in the next 4 years
5. can be contacted

Exclusion Criteria:

1. history of asthma, COPD, lung cancer, active pulmonary tuberculosis, bronchiectasis, diffuse lung disease (interstitial pneumonia, pulmonary sarcoidosis, occupational lung disease, sarcoidosis et al) and pleural disease;
2. history of lobectomy and / or lung transplantation;
3. predicted life expectancy less than 3 years;
4. history of severe psychiatric illnesses, mental disorders, neurological disorders, malignant tumors, chronic liver disease, heart failure, autoimmune diseases, chronic kidney disease;
5. Alcoholism, drug abuse or abuse of toxic solvents;
6. Cannot finish long term follow-up or poor compliance;
7. Do not provide consent

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 10,000 subjects aged 40～75 without history of lung disease will be recruited and followed for 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 10385 (Actual)
Dates: Start 2018-03-03 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-10-09 (Actual)

PRIMARY OUTCOMES:
The incidence of COPD in the second and fourth year and the association between incidence of COPD and rapid decline of FEV1. | 4 years
  FEV1/FVC(forced vital capacity)<70% (after bronchial dilation test);Detect the decline of FEV1(%)by Vitalograph COPD6.

SECONDARY OUTCOMES:
The association between incidence of COPD and the air pollution level in different provinces in China. | 4 years
  Record data of air pollution in different provinces in China from the environmental monitoring website. And analyze the correlation between the COPD incidence and air pollution level.
The association between incidence of COPD and different comorbidity condition, such as metabolic syndrome, cardiovascular disease. | 4 years
  Record comorbidity condition data of human subjects, and then analyze the correlation between the COPD incidence and different comorbidity condition.
The mean decline rate of FEV1 | 4 years
  Monitor pulmonary function decline in the second and the fourth year, then calculate the mean decline value.
The association between decline rate of FEV1 and air pollution level | 4 years
  Record data of air pollution in different provinces in China from the environmental monitoring website. And analyze the correlation between the decline rate of FEV1 and air pollution level.
The correlation between the incidence of COPD and serum IL-6 level. | 4 years
  Detect the serum IL-6 levels(ng/L), then analyze the correlation between the IL-6 levels and COPD incidence.
The correlation between the incidence of COPD and serum hs-CRP level. | 4 years
  Detect the serum hs-CRP levels(ng/L), then analyze the correlation between the hs-CRP levels and COPD incidence.
The association between the pH value of EBC and COPD incidence. | 4 years
  Detect the EBC pH value, then analyze the correlation between the EBC pH value and COPD incidence.
The association between serum miR-23a level and COPD incidence. | 4 years
  Detect the serum miR-23a level, then analyze the correlation between serum miR-23a level and COPD incidence.
The association between incidence of COPD and other factors. | 4 years
  The association between incidence of COPD and other factors (smoking habit, biomass exposure history, eating habit and incoming class).The incidence of COPD in the second and fourth year and the association between incidence of COPD and other factors (smoking habit(has or does not, if has: accumulative total smoking amount), biomass exposure history(yes or no), eating habit(light or greasy) and incoming class(family income per capita >¥4500, or not)).

CONTACTS AND LOCATIONS:
Overall Officials: Guangfa Wang, MD, Study Chair — Peking University First Hospital
Locations (10):
- China (10):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The First Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Shandong Provincial Hospital Affiliated to Shandong University, Jinan, Shandong
  - The First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang X, Liao J, Zhu S, Zhang C, Ma X, Zhang C, Wang Y, Sun K, Wang G. Association of high-sensitivity CRP and FEV1%pred: a study on non-pulmonary disease in a population in Beijing, China. BMJ Open Respir Res. 2024 Mar 13;11(1):e001699. doi: 10.1136/bmjresp-2023-001699. PMID 38479820
- [Derived] Ma X, Zhang C, Wang Y, Yu K, Jin Z, Zhang C, Ma J, Liao J, Wang G. Correlation of morning dry mouth with clinical features of OSA in a community population: a cross-sectional study. Postgrad Med. 2024 Jan;136(1):30-35. doi: 10.1080/00325481.2024.2303972. Epub 2024 Jan 14. PMID 38197225
- [Derived] Wei S, Liao J, Xue T, Yu K, Fu X, Wang R, Dang X, Zhang C, Qiao H, Jiang S, Xiao J, Dong L, Yin J, Yan X, Jia W, Zhang G, Chen R, Zhou B, Song B, Li J, Yin M, Zhang L, Xie L, Dong S, Sun J, Gao P, Miao B, Li W, He L, Ning Q, Zhao L, Liu H, Cao H, Wang G. Ambient fine particulate matter and allergic symptoms in the middle-aged and elderly population: results from the PIFCOPD study. Respir Res. 2023 May 25;24(1):139. doi: 10.1186/s12931-023-02433-2. PMID 37231445
- [Derived] Wang Y, Liao J, Zhong Y, Zhang C, Li X, Wang G. Predictive Value of Combining Inflammatory Biomarkers and Rapid Decline of FEV1 for COPD in Chinese Population: A Prospective Cohort Study. Int J Chron Obstruct Pulmon Dis. 2019 Dec 5;14:2825-2833. doi: 10.2147/COPD.S223869. eCollection 2019. PMID 31824147